CLINICAL TRIAL: NCT06280794
Title: Efficacy of Laser Acupuncture for Idiopathic Bell's Palsy: a Randomized Controlled Trial
Brief Title: Efficacy of Laser Acupuncture for Idiopathic Bell's Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Laser-Bell-2024
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-02

CONDITIONS: Bell's Palsy
Keywords: Idiopathic facial paralysis; Bell's palsy; Laser acupuncture; photobiomodulation; RCT
MeSH Terms: conditions — Bell Palsy | interventions — Steroids

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Laser acupuncture Group (Experimental): Steroids. Patients in the laser acupuncture group (LA group) received 12 sessions of laser acupuncture (3 times per week). Laser aucpuncture used a class IV Multiwave Locked System (MLS) laser (Mphi laser, ASA Srl, Vicenza, Italy).
  In LA group, we choose 5 acupoints on the affected side. It includes ST2(Si Bai), ST4(Di Cang), ST6(Jia Che), GB14(Yang Bai), GB20(Feng chi). We choose 6 acupoints, including LI4 (He Gu), LI11(Qu Chi), ST36 (Zu San Li), SP6 (San Yin Jiao), KI3 (Tai Xi), LR3 (Tai Chong).
  Laser acupuncture used have wavelength of 808 nm and 905nm, 1.2 W power (808nm is 1 W, 905 nm is 200 mW), continuous mode emission (808 nm) and pulsed mode emission (905 nm), 500 Hz, 50% power level, 50% duty cycle, 8.35 J/cm2 dosimetry, 26.22 J for each point, administered for 3 times per week in the first 2 weeks, and 1500 Hz, 50% power level, 50% duty cycle, 8.35 J/cm2 dosimetry, 26.22 J for each point, in the last 2 weeks, 12 times total treatment.
  Interventions: Device: Laser acupuncture; Drug: Steroids
- Sham laser acupuncture Group (Sham Comparator): Steroids. Patients in the laser acupuncture group (LA group) received 12 sessions of laser acupuncture (3 times per week). Laser aucpuncture used a class IV Multiwave Locked System (MLS) laser (Mphi laser, ASA Srl, Vicenza, Italy).
  In LA group, we choose 5 acupoints on the affected side. It includes ST2(Si Bai), ST4(Di Cang), ST6(Jia Che), GB14(Yang Bai), GB20(Feng chi). We choose 6 acupoints, including LI4 (He Gu), LI11(Qu Chi), ST36 (Zu San Li), SP6 (San Yin Jiao), KI3 (Tai Xi), LR3 (Tai Chong).
  The Sham LA group received the same laser device and the same acupoints. The device showed the same red light but did not emit a laser, administered for 3 times per week in the 4 weeks.
  Interventions: Device: Laser acupuncture; Drug: Steroids
- Control group (Other): Steroids.
  Interventions: Drug: Steroids

INTERVENTIONS:
Device: Laser acupuncture — Patients in the laser acupuncture group (LA group) received 12 sessions of laser acupuncture (3 times per week). Laser aucpuncture used a class IV Multiwave Locked System (MLS) laser (Mphi laser, ASA Srl, Vicenza, Italy).
  In LA group, we choose 5 acupoints on the affected side. It includes ST2(Si Bai), ST4(Di Cang), ST6(Jia Che), GB14(Yang Bai), GB20(Feng chi). We choose 6 acupoints, including LI4 (He Gu), LI11(Qu Chi), ST36 (Zu San Li), SP6 (San Yin Jiao), KI3 (Tai Xi), LR3 (Tai Chong).
  Laser acupuncture used have wavelength of 808 nm and 905nm, 1.2 W power (808nm is 1 W, 905 nm is 200 mW), continuous mode emission (808 nm) and pulsed mode emission (905 nm), 500 Hz, 50% power level, 50% duty cycle, 8.35 J/cm2 dosimetry, 26.22 J for each point, administered for 3 times per week in the first 2 weeks, and 1500 Hz, 50% power level, 50% duty cycle, 8.35 J/cm2 dosimetry, 26.22 J for each point, in the last 2 weeks, 12 times total treatment.
  Arms: Laser acupuncture Group; Sham laser acupuncture Group
Drug: Steroids — Prednisolone as 5 mg tablets (Tianjin Lisheng Pharmaceutical Co., Ltd., China) were given as a single dose of 30 mg daily for the first 3 days; 15 mg daily for the following 3 days; 10 mg daily for the after 3 days; 5 mg daily for the final 3 days, with a total treatment time of 9 days.

SUMMARY:
Objective:

Bell's palsy is characterized by acute, unilateral onset that compromises function and esthetics, exerting a considerable impact on the social, professional, and psychological aspects of the lives of affected individuals. The objective of this study was to determine whether laser acupuncture therapy could relieve symptoms in patients with Bell's palsy in 8 weeks.

Methods:

This study was randomized controlled trial including 360 patients that undergoing Bell's palsy. All the patients received oral Prednisolone. Patients were assigned to the laser acupuncture (LA) group, Sham LA group and control group, with 120 patients in each group. LA group and Sham LA group were received 4 weeks of Laser treatment (3 times per week).

Clinical outcome measure comprised the House-Brackmann grading system, Facial Clinimetric Evaluation Scale (FaCE), Sunnybrook facial grading scale (SBFG), Facial Disability Index (FDI) and Facial Clinimetric Evaluation Scale (FaCE Scale) All the measurements were collected at the baseline, weeks 2, 4, 6, 8, 12 and 24.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients diagnosed with idiopathic Bell's Palsy 2.Patients were eligible if they were graded at House-Brackmann grade (HB) 3 or higher.

Exclusion Criteria:

- 1.Serious mental illness or social problems, and neurological disorders, and systemic diseases, such as malignant tumors, and other serious consumptive diseases.

2. Planning for pregnancy, those in pregnancy, or those who were lactating. 3.Bell's Palsy patients who have a disease course of more than 8 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
House Brackmann Grading System (HB) | Baseline, weeks 2, 4, 6, 8, 12 and 24
  The HB is a physician-rated system based on criteria of resting appearance, facial movements, and synkinesis that categorizes facial function from I (normal) to VI (total paralysis), with options of "Normal", "Mild dysfunction", "Moderate dysfunction", "Moderately severe dysfunction", "Severe dysfunction" or "Total paralysis". The prognoses of grade 3 or higher were abnormal.

SECONDARY OUTCOMES:
Sunnybrook Facial Grading Scale (SB Grading) | Baseline, weeks 2, 4, 6, 8, 12 and 24
  The Sunnybrook Facial Grading Scale was used because of its international recognition and because it allowed a separate classification of the degree of synkinesis. The SB Grading is divided into three subscales of resting symmetry (Eye and Mouth range from 0 to 1, Cheek ranges from 0 to 2), symmetry of voluntary movement (ranges from 1 to 5), and synkinesis (ranges from 0 to 3). The three subscores are used to calculate a composite score (ranges from 0 to 100).
Facial Disability Index (FDI) | Baseline, weeks 2, 4, 6, 8, 12 and 24
  Facial Disability Index (FDI) is a brief, self-report questionnaire of physical disability and psychosocial factors related to facial neuromuscular function. The FDI is a 10-item test that is divided into physical function (ranges from 0 to 5). and social/ well-being function (ranges from 1 to 6) domains. The physical function scores range from -25 (worst) to 100 (best), and the social/wellbeing function scores range from 0 (worst) to 100 (best).
Facial Clinimetric Evaluation Scale (FaCE Scale) | Baseline, weeks 2, 4, 6, 8, 12 and 24
  FaCE is 15-items, self-reported questionnaire that used to assess facial impairment and disability after facial paralysis. It includes six independent domains: social function, facial movement, facial comfort, oral function, eye comfort, and lacrimal control. the total scores range from 0 (worst) to 100 (best).

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing TongRen Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes